CLINICAL TRIAL: NCT02202798
Title: New Devices to Measure the Intracuff Pressure
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00741
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Patients Intubated With a Cuffed Endotracheal Tube
MeSH Terms: interventions — Syringes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Syringe device: Endotracheal tube cuff pressure measured by 2 new syringe devices.
  Interventions: Device: Syringe device

INTERVENTIONS:
Device: Syringe device
  Other Names: Tru-Cuff; AG Cuffill

SUMMARY:
Over the past 5 years, there has been a change in clinical practice with the use of cuffed instead of uncuffed endotracheal tubes in infants and children. Two manufacturing companies have recently introduced syringe-like devices to the market which allow the measurement of the intracuff pressure. This study proposes to prospectively compare the intracuff pressure from these devices with the gold standard technique (manometer).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or younger, undergoing a procedure requiring endotracheal intubation with a cuffed ETT.

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients that are being intubated with a cuffed endotracheal tube prior to surgery.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Cuff pressure | One time in the OR prior to the start of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States